CLINICAL TRIAL: NCT02735590
Title: A Randomized, Partially-blinded, Clinical Trial of Isoniazid and Rifapentine (3HP) Therapy to Prevent Pulmonary Tuberculosis in High-risk Individuals Identified by a Transcriptomic Correlate of Risk
Brief Title: The Correlate of Risk Targeted Intervention Study
Acronym: CORTIS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cape Town (Other)
Collaborators: South African Tuberculosis Vaccine Initiative (Other); Aurum Institute (Other); Centre for the AIDS Programme of Research in South Africa (Network); University of Stellenbosch (Other); London School of Hygiene and Tropical Medicine (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Mark Hatherill, National Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CORTIS-01
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open-label 3HP (Experimental): Participants in the Treatment Arm will receive high dose INH (15mg per kg body weight, rounded up to the nearest 100 mg; maximum dose 900 mg) with Pyridoxine supplementation (25mg), and Rifapentine based on body weight (>32kg - 50kg: 750 mg; >50kg: 900 mg), given weekly as 12 directly observed treatment (DOT) oral doses, ideally with food, over 3 months. Dispensing of IP and Directly Observed Treatment (DOT) field visits in Treatment Arm participants will be performed by staff members not involved in TB symptom screening or investigation. Participants receiving 3HP who develop symptoms of hepatotoxicity will be evaluated by an Investigator.
  Interventions: Drug: Isoniazid; Drug: Rifapentine
- Baseline Screening; Active Surveillance (No Intervention): Adult volunteers living in TB hyperendemic communities of South Africa will be consented and screened. Individuals with HIV infection and conditions likely to affect the performance of the COR assay, or the safety and/or efficacy of the 3HP investigational regimen, will not be enrolled. Active surveillance for TB disease (Observation Arm), including regular symptom screening and symptom-targeted TB investigation (all participants) will be conducted on this Arm.

INTERVENTIONS:
Drug: Isoniazid — Participants in the Treatment Arm will receive high dose Isoniazid - 15mg per kg body weight, rounded up to the nearest 100 mg; maximum dose 900 mg with Pyridoxine supplementation (25mg).
  Arms: Open-label 3HP
Drug: Rifapentine — Rifapentine based on body weight (>32kg - 50kg: 750 mg; >50kg: 900 mg), given weekly as 12 directly observed treatment (DOT) oral doses, ideally with food, over 3 months.
  Arms: Open-label 3HP

SUMMARY:
Effective tuberculosis (TB) control requires that people who progress from latent Mycobacterium tuberculosis (MTB) infection (LTBI) to TB disease are identified and treated before they infect others. A prognostic correlate of risk (COR), based on messenger ribonucleic acid (mRNA) expression signatures, which prospectively discriminates between TB cases and healthy controls, has been constructed and validated. Based on published microarray case-control datasets, the COR has 87% diagnostic sensitivity and 97% specificity for prevalent TB disease; and in two nested case-control studies, 70% prognostic sensitivity and 84% specificity for incident TB disease occurring within one year of sampling (HIV uninfected persons). Diagnostic and prognostic performance of the COR has not yet been tested in a prospective cohort.

COR+ status is not directly associated with LTBI; and may, or may not, be amenable to preventive therapy. Although effective in the short-term, preventive therapy is not recommended for treatment of LTBI in HIV uninfected adults living in high TB burden countries, due to rapid loss of protection; and treatment burden. A 3-month, 12-dose, once-weekly preventive therapy regimen of high dose Isoniazid (INH) and Rifapentine (3HP) has been recommended as equivalent to 6 months of daily INH for treatment of LTBI in low TB burden countries by the World Health Organization (WHO).

A 'screen & treat' strategy, based on serial mass campaigns to provide targeted, short-course preventive therapy only to COR+ persons at highest risk of TB disease, may offer the solution for durable, community-wide protection in high TB burden countries. The efficacy of 3HP for prevention of incident TB disease in COR+ persons has not yet been tested in a clinical trial.

Primary Aims

1. Test whether preventive therapy (3HP) reduces the rate of incident TB disease, compared to standard of care (active surveillance), in COR+ persons.
2. Test whether COR status differentiates persons with cumulative prevalent or incident TB disease from persons without TB disease.

Secondary Aims

1. Estimate whether COR status differentiates persons at high risk for incident TB disease from persons at low risk for incident TB disease
2. Compare prognostic performance of the COR for incident TB disease with Interferon-gamma release assay (IGRA).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged ≥18 and <60 years
3. Known COR status (- or +)
4. Known HIV status
5. Women of child-bearing potential who are not surgically sterilized must agree to practice adequate contraception (barrier method or non-hormonal intrauterine device, alone or in addition to systemic hormonal contraceptive method) or abstain from heterosexual intercourse during the first 3 months on study.
6. Likely to remain in follow-up and adhere to protocol requirements

Exclusion Criteria:

1. HIV infection
2. Pregnant or lactating
3. Diagnosed with TB disease within last 3 years
4. Household exposure to a TB patient with known multi-drug resistant (MDR-) TB disease within last 3 years
5. Body weight <40kg
6. Known allergy to INH or Rifamycins
7. Receiving antiarrhythmic, antidepressant, antipsychotic, antihypertensive, anticonvulsant, anticoagulant, or (inhaled or oral) corticosteroid therapy
8. Any medical, surgical, or other condition, including but not limited to known diabetes mellitus (requiring oral or injectable therapy), liver disease, porphyria, peripheral neuropathy, epilepsy, psychosis, or alcoholism, that in the opinion of the Investigator is likely to interfere with COR performance; safety and efficacy of the investigational products (IP); or adherence to protocol requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2927 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy | 15 months
  Treatment efficacy (TE) will be evaluated by comparing the incidence of endpoint-defined TB disease over 15 months in treated COR+ versus untreated COR+ participants.
Performance of COR | 15 months
  The performance of the COR will be evaluated by comparing the cumulative incidence of endpoint-defined TB disease over 15 months in untreated COR+ versus untreated COR- participants

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, MD, FCP (SA), Principal Investigator — South African Tuberculosis Vaccine Initiative
Locations (5):
- South Africa (5):
  - Centre for the Aids Programme of Research in South Africa (CAPRISA), Durban, KwaZulu-Natal
  - Aurum Institute, Klerksdorp, North West
  - Aurum Institute, Rustenburg, North West
  - Stellenbosch Immunology Research Group, Cape Town, Western Cape
  - South African Tuberculosis Vaccine Initiative (SATVI), Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Publications

REFERENCES:
- [Derived] Scriba TJ, Fiore-Gartland A, Penn-Nicholson A, Mulenga H, Kimbung Mbandi S, Borate B, Mendelsohn SC, Hadley K, Hikuam C, Kaskar M, Musvosvi M, Bilek N, Self S, Sumner T, White RG, Erasmus M, Jaxa L, Raphela R, Innes C, Brumskine W, Hiemstra A, Malherbe ST, Hassan-Moosa R, Tameris M, Walzl G, Naidoo K, Churchyard G, Hatherill M; CORTIS-01 Study Team. Biomarker-guided tuberculosis preventive therapy (CORTIS): a randomised controlled trial. Lancet Infect Dis. 2021 Mar;21(3):354-365. doi: 10.1016/S1473-3099(20)30914-2. Epub 2021 Jan 25. PMID 33508224